CLINICAL TRIAL: NCT07378852
Title: Integrated Study on Gut Microbiota, Immune Indicators, and Trace Elements in Children With Respiratory Tract Infections
Status: Not yet recruiting | Type: Observational
Sponsor: Min-Tze LIONG (Other)
Collaborators: The 940th Hospital of the Joint Logistic Support Force of the Chinese People's Liberation Army (Unknown)
Responsible Party: Sponsor-Investigator, Min-Tze LIONG, Prof., Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Other Study IDs: 2024KY22213
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Respiratory
Keywords: children; respiratory; gut microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mycoplasma pneumoniae pneumonia (MPP) group: Children with Mycoplasma pneumoniae pneumonia
- Non-mycoplasma acute respiratory tract infection (NMP) group: Children with acute respiratory tract infection without Mycoplasma pneumoniae
- Recurrent respiratory tract infections (RRTIs) group: Children with recurrent respiratory tract infections
- Healthy control group: Healthy children without any respiratory disease

SUMMARY:
This observational study aims to investigate the characteristics of gut microbiota and their associations with immune and nutritional indicators in children with different respiratory health statuses. A total of 120 children will be enrolled and categorized into four groups: children with Mycoplasma pneumoniae pneumonia (MPP), children with acute respiratory tract infections without Mycoplasma pneumoniae (NMP), children with recurrent respiratory tract infections (RRTIs), and healthy controls. By comparing gut microbiota composition and diversity, as well as immune- and nutrition-related indicators across groups, this study seeks to clarify the potential role of intestinal dysbiosis and host immune-nutritional interactions in the pathogenesis and clinical manifestations of pediatric respiratory tract infections.

DETAILED DESCRIPTION:
Respiratory tract infections remain one of the leading causes of morbidity in children. Among them, Mycoplasma pneumoniae pneumonia (MPP) and recurrent respiratory tract infections (RRTIs) represent two clinically important yet mechanistically heterogeneous disease patterns. The former is characterized by acute inflammatory responses and immune dysregulation, whereas the latter reflects long-term susceptibility, immune imbalance, and repeated infectious episodes.

In recent years, the gut microbiota has been recognized as a critical regulator of systemic immunity through the gut-lung axis. Alterations in intestinal microbial composition have been implicated in respiratory infection susceptibility, inflammatory regulation, and immune maturation in children. In parallel, essential trace elements such as zinc and iron play indispensable roles in maintaining mucosal barrier integrity, immune function, and microbial homeostasis. However, integrated evidence linking gut microbiota characteristics, immune-related indicators, and trace element status across different pediatric respiratory disease phenotypes remains limited.

Therefore, this study adopts a prospective observational case-control design. From November 2024 to June 2026, a total of 120 children aged 3-14 years will be enrolled and divided equally into four groups (30 participants per group), namely mycoplasma pneumoniae pneumonia (MPP) group, non-mycoplasma acute respiratory tract infection (NMP) group, recurrent respiratory tract infections (RRTIs) group, and healthy control group.

Clinical information and fecal samples will be collected according to standardized procedures. Gut microbiota composition and diversity will be analyzed using fecal samples, while immune- and nutrition-related indicators will be assessed in accordance with established laboratory protocols. Comparative and correlation analyses will be conducted to explore disease-specific microbial and host response patterns.

This integrated study aims to provide a comprehensive biological basis for understanding pediatric respiratory infections and to support future strategies involving microbiota modulation, nutritional intervention, and immune regulation.

ELIGIBILITY:
Inclusion Criteria

1. Aged 3-14 years;
2. Good compliance and complete clinical data;
3. Guardians are informed and sign written consent;
4. MPP group: meets diagnostic criteria of Guidelines for Diagnosis and Treatment of Mycoplasma Pneumoniae Pneumonia in Children (2023 Edition);
5. NMP group: acute respiratory tract infection with negative MP-DNA/RNA;
6. RRTIs group: meets diagnostic criteria of Clinical Diagnosis and Treatment Pathway for Recurrent Respiratory Tract Infections in Children (2022 Edition);
7. Healthy controls: no respiratory infection history within the past month.

Exclusion Criteria

1. Other infectious diseases (e.g., measles, pertussis, tuberculosis);
2. Congenital heart disease, immunodeficiency, or major organ dysfunction;
3. Use of antibiotics, probiotics, immunomodulators, hormones, or microecological preparations within the past 15-30 days;
4. Unqualified biological samples or incomplete laboratory data.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children from all cohorts will be recruited from the pediatric clinics of the 940th Hospital of the Joint Logistics Support Force of the Chinese People's Liberation Army
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Microbiota profiles of fecal samples in all children cohorts as assessed via metagenomics sequencing | Day-1
  Differences in microbiota abundance in fecal sample of children with respiratory diseases compared to healthy cohort

SECONDARY OUTCOMES:
Respiratory symptoms duration and frequency in all children cohorts as assessed using questionnaire | Day-1
  Changes in duration and frequency of respiratory illnesses symptoms from children with respiratory diseases and healthy cohort, via the use of standard clinical assessment questionnaire, scale 0-3 where higher scores indicate more severe symptoms.
Gastrointestinal symptoms duration and frequency in all children cohorts as assessed using questionnaire | Day-1
  Changes in duration and frequency of gastrointestinal illnesses symptoms from children with respiratory diseases and healthy cohort, via the use of standard clinical assessment questionnaire, scale 0-3 where higher scores indicate more severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Yongli Dai, MD., Principal Investigator — The 940th Hospital of the Joint Logistic Support Force of the Chinese People's Liberation Army
Locations (2):
- The 940th Hospital of the Joint Logistic Support Force of the Chinese People's Liberation Army, Lanzhou, Gansu, China
- Universiti Sains Malaysia, Pulau Pinang, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No